CLINICAL TRIAL: NCT03364764
Title: Sirolimus Treatment for Refractory Pure Red Cell Aplasia, a Prospective Study
Brief Title: Sirolimus Treatment for Refractory PRCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bing Han (Other)
Responsible Party: Sponsor-Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRCA-1
Record Dates: First submitted 2017-11-21; First posted 2017-12-07 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2020-06

CONDITIONS: Pure Red Cell Aplasia
Keywords: sirolimus; refractory pure red cell aplasia; prospective study
MeSH Terms: conditions — Red-Cell Aplasia, Pure | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- efficiency of sirolimus on PRCA (Experimental): A prospective research of the sirolimus efficiency on refractory PRCA patients On refractory PRCA patients, sirolimus was tried. Dosage: 2mg QD for the first day, then 1 mg QD. Medication time should last at least 6 months.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — On refractory PRCA patients, sirolimus was tried. Dosage: 2mg QD for the first day, then 1 mg QD. Medication time should last at least 6 months.
  Other Names: Sirolimus Tablets

SUMMARY:
Pure red cell aplasia (PRCA) is a kind of anemia characterized by severe reticulocytopenia and obvious bone marrow erythroblastic cells decreased. Cyclosporine and /or steroids are the first line therapy but some patients were refractory or intolerance to the treatment. The effects of the second line therapy are also not satisfactory and sometimes not available. The investigators aim to explore the efficacy and side-effect of sirolimus for refractory PRCA.

DETAILED DESCRIPTION:
Pure red cell aplasia (PRCA) is a rare normocytic normochromic anemia with reticulocytopenia, characterized by a reduction of erythroid precursors from the bone marrow, could be divided into congenital and acquired PRCA according to pathogenesis. Congenital PRCA, also known as Diamond-Blackfan syndrome, has been associated with pathogenic variant in GATA1 and TSR2 and gene encode ribosomal proteins. Acquired PRCA can be a primary disease which is usually mediated by immunology, or secondary to other diseases, such as lymphoproliferative diseases, autoimmune diseases, thymoma, infection, or drugs. The first line therapy of acquired PRCA is Cyclosporine A and steroids, the second line therapy are anti-CD20, ATG, immunosuppressive drugs like cyclophosphamide, bone marrow transplantation. Unfortunately, some patients did not response or tolerate the above treatments.

Sirolimus (rapamycin) is an agent produced by the bacterium Streptomyces hygroscopicus, inhibits the mammalian target of rapamycin (mTOR). mTOR is a serine/threonine kinase that regulates cell growth, proliferation, metabolism and survival in eukaryotic cells, and is identified as two interacting complex, mTORC1 and mTORC2. Sirolimus primarily inhibits mTORC1, has been approved for prevent organ transplant rejection, especially in renal transplantation, sirolimus also promises to treat autoimmune, degenerative and hyperproliferative disorders. Recently, sirolimus has been reported to be effective and well tolerated for many immune-mediated cytopenias, such as autoimmune lymphoproliferative syndrome, immune thrombocytopenia, EVANS syndrome, etc. However, due to the rare occurrence of PRCA and good response rate to cyclosporine, there are very few studies of sirolimus on refractory PRCA so far.

In this study, It is anticipate to evaluate the effect of sirolimus on 30 patients with refractory PRCA, the side-effects was documented and plasma concentration of sirolimus will be monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory pure red cell aplasia.
2. Excluding other diseases which might cause hematological abnormalities.
3. No response or intolerant to first and second line therapies.
4. 18-80 years old.
5. All subjects must: agree not to donate blood or be counseled about pregnancy precautions and risks of fetal exposure.
6. Written informed consent.

Exclusion Criteria:

1. NOT refractory pure red cell anemia.
2. Response and well tolerate to first or second line therapy.
3. Patients who are under 18-year-old or over 80-year-old.
4. Pregnant or lactating.
5. Patients unwilling to or unable to comply with the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | 6 months
  Hemoglobin level in g/L

SECONDARY OUTCOMES:
Hemoglobin level | 2 years
  Hemoglobin level in g/L

CONTACTS AND LOCATIONS:
Overall Officials: Bing B Han, PhD., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bride KL, Vincent T, Smith-Whitley K, Lambert MP, Bleesing JJ, Seif AE, Manno CS, Casper J, Grupp SA, Teachey DT. Sirolimus is effective in relapsed/refractory autoimmune cytopenias: results of a prospective multi-institutional trial. Blood. 2016 Jan 7;127(1):17-28. doi: 10.1182/blood-2015-07-657981. Epub 2015 Oct 26. PMID 26504182
- [Result] Li J, Wang Z, Dai L, Cao L, Su J, Zhu M, Yu Z, Bai X, Ruan C. Effects of rapamycin combined with low dose prednisone in patients with chronic immune thrombocytopenia. Clin Dev Immunol. 2013;2013:548085. doi: 10.1155/2013/548085. Epub 2013 Dec 2. PMID 24363761
- [Result] Means RT Jr. Pure red cell aplasia. Blood. 2016 Nov 24;128(21):2504-2509. doi: 10.1182/blood-2016-05-717140. PMID 27881371
- [Result] Teachey DT, Greiner R, Seif A, Attiyeh E, Bleesing J, Choi J, Manno C, Rappaport E, Schwabe D, Sheen C, Sullivan KE, Zhuang H, Wechsler DS, Grupp SA. Treatment with sirolimus results in complete responses in patients with autoimmune lymphoproliferative syndrome. Br J Haematol. 2009 Apr;145(1):101-6. doi: 10.1111/j.1365-2141.2009.07595.x. Epub 2009 Feb 4. PMID 19208097